CLINICAL TRIAL: NCT02268643
Title: Ultrasound-based Breast Cancer Screening in Chinese Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Qiang SUN, Director, Peking Union Medical College Hospital
Other Study IDs: PUMCH-breast-screening 2
Record Dates: First submitted 2014-09-29; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; screening; ultrasound; risk model
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- group 1: ultrasound plus clinical breast examination
  Interventions: Other: ultrasound plus clinical breast examination

INTERVENTIONS:
Other: ultrasound plus clinical breast examination — all the participants will be required to fill risk factor questionaires and then be screened with ultrasound plus physical examination every year

SUMMARY:
In the present study, the investigators will screen breast cancer of the Chinese women based on ultrasound and aim to compare the risk evaluation model of PUMCH model which was established by our previous work with other risk models.

DETAILED DESCRIPTION:
Early detection of breast cancer through screening has been a common practice in the United States and several European countries for decades. It is effective in reducing the mortality of breast cancer and improving the postoperative quality of life of patients. Mammography has been the standard imaging method for the screening, however, our previous study has shown that ultrasound is more sensitive and less expensive than mammography. In the present study, the investigators will screen breast cancer of the Chinese women based on ultrasound and aim to evaluate the risk model (PUMCH model) which was established by our previous work.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent；
* residence from community or working units

Exclusion Criteria:

* pregnancy；
* lactation；
* known metastatic cancer；
* signs or symptoms of breast disease；
* presence of breast implants, breast surgery within prior 12 months；
* had mammography or ultrasound exam within prior 12 months
* males.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy women without breast-related symptoms
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
number of cancer detected in the high-risk group | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sun Qiang, MD, Study Chair — PUMCH
Locations (16):
- China (16):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing ChaoYang Hospital affiliated to the Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital affiliated to Ministry of Health, Beijing, Beijing Municipality
  - First Hospital affiliated to Peking University, Beijing, Beijing Municipality
  - Southwest Hospital affiliated to the Third Military Medical University, Chongqing, Chongqing Municipality
  - ShanXi Traditional Medicine Hospital, Taiyuan, Shanxi
  - The Cancer Hospital affiliated to Tianjin Medical University, Tianjin, Tianjin Municipality
  - Chifeng Baoshan Hospital, Chifeng
  - First Affiliated Hospital of Chongqing Medical University, Chongqing
  - First People's Hospital of Honghe State, Mengzi
  - Ordos Central Hospital, Ordos
  - Qingdao Municipal Hospital, Qingdao
  - First Affiliated Hospital of China Medical University, Shenyang
  - Hospital of Xinjiang Production and Construction Corps, Ürümqi
  - Third Hospital of Xingtai, Xingtai
  - Yingshan Maternal and Child Health Hospital, Yingshan